CLINICAL TRIAL: NCT05571904
Title: The Comparison of Thick Split-thickness Skin Graft Versus Thin Split-thickness Skin Graft in the Reconstruction of the Donor Site
Brief Title: The Comparison of Thick Split-thickness Skin Graft Versus Thin Split-thickness Skin Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, YinWu, attending doctor of Department of Burn and Plastic Surgery,Nanjing First Hospital, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20220701-08
Record Dates: First submitted 2022-10-06; First posted 2022-10-07 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Reconstruction
Keywords: donor site; thick split-thickness skin graft; thin split-thickness skin graft; reconstruction

STUDY DESIGN:
Intervention Model Description: (1) Patients had skin defects at functional sites or joint sites; (2) Patients aged 20-80 years; (3) The lateral thighs were chosen as the donor sites.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the thick STSG group (Experimental): For the patients in the thick STSG group, the surgeons harvested thick STSGs which were larger than recipient sites. The extra skin was punctured and stretched to cover the donor site (the novel technique).
  Interventions: Procedure: thick STSG; thin STSG
- the thin STSG group (Active Comparator): For the patients in the thin STSG group, the surgeons harvested thick STSGs of the size of recipient sites. Their donor sites were covered with thin STSGs which were harvested from other parts of the patients.
  Interventions: Procedure: thick STSG; thin STSG

INTERVENTIONS:
Procedure: thick STSG; thin STSG — For all the patients, thick STSGs (at a depth of 0.7 mm) were harvested from the upper lateral thighs to repair skin defects at functional sites or joint sites. For patients in the thick STSG group, the surgeons harvested a larger size of thick STSGs than the size of recipient sites. The size of the donor site was 150% - 200% of the size of the recipient site. Part of the thick STSG was grafted onto the recipient site. Subsequently, the leftover skin was punctured (in 1.5:1 mesh ratio) and stretched to obtain expansion. The donor site was covered by the leftover skin completely. In other words, the donor site was reconstructed by resurfacing the large sheet of thick STSG in situ.
  For patients in the thin STSG group, the surgeons harvested thick STSGs of the size of recipient sites. Their donor sites were covered with a large sheet of thin STSGs (at a depth of 0.4 mm) which were harvested from other parts of the patients.

SUMMARY:
In clinical settings, split-thickness skin graft (STSG) remain the gold standard for covering large skin defects. However, STSGs usually bring complications to the donor sites. The study objective was to compare the efficacy of thick split-thickness skin graft versus thin split-thickness skin graft in the reconstruction of the donor site.

DETAILED DESCRIPTION:
All patients were randomly divided into two groups. For the patients in the thick STSG group, the surgeons harvested thick STSGs which were larger than recipient sites. The extra skin was punctured and stretched to cover the donor site (the novel technique). For the patients in the thin STSG group, the surgeons harvested thick STSGs of the size of recipient sites. Their donor sites were covered with thin STSGs which were harvested from other parts of the patients. The 36-item short form health survey (SF-36) scores, pain scores, pruritus scores, scar scores and rates of complications were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had skin defects at functional sites or joint sites.
2. Patients aged 20-80 years.
3. The lateral thighs were chosen as the donor sites.

Exclusion Criteria:

1. Patients who were unable to complete the follow-up.
2. Pregnant or nursing mothers were not included.
3. Patients had an alternative source of pain other than surgical sites.
4. Patients with organ dysfunctions (heart failure, respiratory failure, liver dysfunction, renal impairment or intestinal failure), or cancers.
5. Patients with autoimmune diseases (rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, Sjogren's syndrome, connective tissues disease or systemic vasculitis) were not included.
6. Patients who had medications (such as corticosteroids, immunosuppressive agents or chemotherapy) within six months were not included.
7. Other reasons.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
healing time of the donor sites | 2 months post surgery
  The complete healing time of the donor sites was defined as the day when 100% epithelialization was achieved,

SECONDARY OUTCOMES:
life quality (36-item short form health survey scores) | Prior to surgery or at 6 months post-surgery
  The life quality of patients was evaluated by the 36-item short form health survey (SF-36) scores (including General Health scores, Mental Health scores, Social Function scores, and Vitality scores). The minimum value is 0. The maximum value is 100. The higher score means a better outcome.
pains scores (Visual Analogue Scales) | on Day 1 and Day 7 postoperatively
  The degrees of pain at the donor sites were evaluated by the Visual Analogue Scales. Patients were asked to score levels of pain (0 = no pain, 5 = worst pain) using Visual Analogue Scales. The higher score means a worse outcome.
pruritus scores | at 3 months and at 6 months post-surgery
  The degrees of pruritus at the donor sites were measured by scores (1 = never or occasional itches, 2 = itches do not disturb sleep, 3= itches disturb sleep). The higher score means a worse outcome.
scars scores ( Vancouver Scar Scales ) | at 3 months and 6 months post-surgery
  The scar formation at the donor sites were evaluated with the Vancouver Scar Scales (from 0 to 15, 0 = best and 15 = worst) in terms of pigmentation, vascularity, pliability and height. The higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Wu, phD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, Iinformed Consent Form will be shared on the website:http://www.stats.gov.cn/tjsj/
Supporting Information: Study Protocol, ICF, CSR
Time Frame: December,31,2023
Access Criteria: no limits
URL: http://www.stats.gov.cn/tjsj/

REFERENCES:
- [Background] Bian Y, Sun C, Zhang X, Li Y, Li W, Lv X, Li J, Jiang L, Li J, Feng J, Li XY. Wound-healing improvement by resurfacing split-thickness skin donor sites with thin split-thickness grafting. Burns. 2016 Feb;42(1):123-130. doi: 10.1016/j.burns.2015.07.008. Epub 2015 Nov 23. PMID 26615713
- See also: Pubmed — https://pubmed.ncbi.nlm.nih.gov/26615713/